CLINICAL TRIAL: NCT02834273
Title: Impact of Patient Education Following a Stroke on Knowledge of Risk Factors, Stroke Warning Signs and What to do in Cases of Stroke
Brief Title: Patient Education Following a Stroke
Acronym: EPIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2013/18
Record Dates: First submitted 2016-06-20; First posted 2016-07-15 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Therapeutic Workshop (Experimental): Therapeutic Workshop (patients following therapeutic education workshops during their hospitalization)
  Interventions: Behavioral: stroke education workshops
- Usual care (No Intervention)

INTERVENTIONS:
Behavioral: stroke education workshops
  Arms: Therapeutic Workshop

SUMMARY:
The rapid diagnosis and treatment of acute ischemic stroke are critical in the reduction of morbidity, disability and stroke associated mortality Under-education about stroke may prevent people from recognizing symptoms early enough to seek immediate care.

The studies reported on stroke patients managed in stroke center have shown that 39-42% of patients could not name any symptoms of stroke and 36% to 43% no risk factor of stroke.

The stroke patients are therefore a population at high risk for neurological events and cardiac vascular recurrence. However, no studies have evaluated the interest of the development of therapeutic workshops in stroke unit to educate patients about symptoms suggestive of stroke, risk factors and what to do in cases of stroke.

Investigators assume that the setting up of a therapeutic education workshop in the stroke unit may allow a better understanding of the symptoms, risk factors and what to do following stroke. So there is a direct benefit to the patient represented by a better knowledge of stroke (warning signs, risk factors, what to do), improved treatment compliance and reduced risk of recurrence.

More generally, there is a real benefit to promote these messages to the public through the patient and his relatives

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years.
* Diagnosis of ischemic stroke;
* Patients with back home or shorter rehabilitation;
* Patients affiliated to a social security scheme;
* Patients who consented to participate in writing.

Exclusion Criteria:

* Patients with cognitive disorders, vigilance, aphasia.
* Patients institutionalized.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2013-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Questionnaire EPIC score | 3 months
  The questionnaire score will concern knowledge of stroke risk factors, alert symptoms and what to do :
  1 point by quoted risk factor, 2 points by quoted symptom and 3 by quoted conduct

SECONDARY OUTCOMES:
Blood pressure | 12 months
LDL-C | 12 months
Body Mass Index | 12 months
Smoking intoxication | 12 months
Recurrent stroke | 12 months
Compliance to treatments | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Lapergue, MD PhD, Principal Investigator — Hopital Foch
Locations (1):
- Hopital Foch, Suresnes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Crocker TF, Brown L, Lam N, Wray F, Knapp P, Forster A. Information provision for stroke survivors and their carers. Cochrane Database Syst Rev. 2021 Nov 23;11(11):CD001919. doi: 10.1002/14651858.CD001919.pub4. PMID 34813082